CLINICAL TRIAL: NCT06586840
Title: The Effect of Adding an IPACK Block to the Adductor Canal Block on Postoperative Pain and Hospital Stay in Patients Undergoing Total Knee Arthroplasty Surgery
Brief Title: The Effect of Adding an IPACK Block to the Adductor Canal Block on Total Knee Arthroplasty Surgery
Status: Recruiting | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, MURAT DEMİRCİOGLU, doctor, Aydin Adnan Menderes University
Other Study IDs: 2023/07/01
Record Dates: First submitted 2024-08-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Pain, Acute
Keywords: adductor canal block; knee arthroplasty; ipack
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adductor Canal Block: For Group I, after patients are placed in the supine position, a linear ultrasound probe (13-6 MHz) will be used to identify the superficial femoral artery in the short axis, lateral to the Sartorius muscle, and anterior to the adductor magnus muscle in the adductor canal. A 22-gauge × 100 mm needle (Braun® Stimuplex) will be inserted in-plane laterally to medially under sterile conditions, and 20 mL of 0.5% bupivacaine will be injected after negative aspiration.
  Interventions: Other: rescue analgesia; Procedure: Adductor Canal Block
- Adding an IPACK Block to the Adductor Canal Block: For Group II, 20 mL of 0.25% bupivacaine will be injected into the Adductor Canal after spinal anesthesia. With the knee flexed, a convex probe (3.5-6 MHz) will be placed in the popliteal region to identify the popliteal artery in the short axis. The ultrasound probe will be moved distally after the common peroneal and tibial nerves are identified. The probe will be gradually moved towards the popliteal fossa until the popliteal vessels are identified superficially. The ultrasound probe will be moved to the level where the femoral condyles merge with the femoral shaft. The popliteal artery, tibial and peroneal nerves will be visualized to identify the space between the femur and the popliteal artery. In the area known as iPACK, a 22-gauge × 100 mm needle (Braun® Stimuplex) will be inserted in-plane laterally to medially, and 20 mL of 0.25% bupivacaine will be injected after negative aspiration.
  Interventions: Other: rescue analgesia; Procedure: Adding an IPACK Block to the Adductor Canal Block

INTERVENTIONS:
Other: rescue analgesia — . If NRS is 4 or higher in the postoperative recovery room, 100 mg of intravenous tramadol will be administered as rescue analgesia
Procedure: Adductor Canal Block — For Group I, after patients are placed in the supine position, a linear ultrasound probe (13-6 MHz) will be used to identify the superficial femoral artery in the short axis, lateral to the Sartorius muscle, and anterior to the adductor magnus muscle in the adductor canal. A 22-gauge × 100 mm needle (Braun® Stimuplex) will be inserted in-plane laterally to medially under sterile conditions, and 20 mL of 0.5% bupivacaine will be injected after negative aspiration.
  Groups: Adductor Canal Block
Procedure: Adding an IPACK Block to the Adductor Canal Block — For Group II, 20 mL of 0.25% bupivacaine will be injected into the Adductor Canal after spinal anesthesia. With the knee flexed, a convex probe (3.5-6 MHz) will be placed in the popliteal region to identify the popliteal artery in the short axis. The ultrasound probe will be moved distally after the common peroneal and tibial nerves are identified. The probe will be gradually moved towards the popliteal fossa until the popliteal vessels are identified superficially. The ultrasound probe will be moved to the level where the femoral condyles merge with the femoral shaft. The popliteal artery, tibial and peroneal nerves will be visualized to identify the space between the femur and the popliteal artery. In the area known as iPACK, a 22-gauge × 100 mm needle (Braun® Stimuplex) will be inserted in-plane laterally to medially, and 20 mL of 0.25% bupivacaine will be injected after negative aspiration.
  Groups: Adding an IPACK Block to the Adductor Canal Block

SUMMARY:
Total knee arthroplasty (TKA) is a frequently performed major orthopedic surgery, where most patients experience severe postoperative pain. Pain-related delays in patient mobilization can lead to thromboembolism, deep vein thrombosis, surgical site infection, and increased risk of hospital-acquired infections due to prolonged hospital stay. Optimal postoperative knee analgesia is crucial not only for patient comfort and satisfaction but also for accelerating mobilization, functional recovery, and discharge from the hospital. To facilitate early ambulation and superior performance, multimodal analgesia and motor-sparing blocks are increasingly utilized

DETAILED DESCRIPTION:
In total knee arthroplasty, a pain management method that preserves motor strength is increasingly accepted as part of the perioperative rehabilitation protocol. Although peripheral nerve blocks like the femoral nerve block (FNB) can cause significant loss of quadriceps muscle strength and delayed rehabilitation due to the risk of patient falls, growing evidence supports the use of the Total knee arthroplasty (TKA) is a frequently performed major orthopedic surgery, where most patients experience severe postoperative pain. Pain-related delays in patient mobilization can lead to thromboembolism, deep vein thrombosis, surgical site infection, and increased risk of hospital-acquired infections due to prolonged hospital stay. Optimal postoperative knee analgesia is crucial not only for patient comfort and satisfaction but also for accelerating mobilization, functional recovery, and discharge from the hospital. To facilitate early ambulation and superior performance, multimodal analgesia and motor-sparing blocks are increasingly utilized.

Regional anesthesia techniques are among the most effective methods for postoperative analgesia. Peripheral nerve blocks, a type of regional anesthesia, provide ideal postoperative analgesia due to their ability to offer effective analgesia, reduce opioid requirements and associated side effects, and facilitate recovery by effectively managing dynamic pain.

The innervation of the knee joint is supplied by branches from the femoral nerve, obturator nerve, common peroneal nerve, and tibial nerve, which originate from the lumbar and sacral plexuses responsible for lower extremity innervation.

adductor canal block (ACB) in total knee arthroplasty patients for minimal motor involvement or purely sensory block.

The adductor canal block (ACB) is a predominantly sensory nerve block that includes the saphenous nerve, the nerve to the vastus medialis muscle, and the articular branches of the obturator nerve. When performed successfully, it provides analgesia similar to the femoral nerve block without significant motor loss in the thigh. It is primarily used for lower extremity surgeries such as total knee arthroplasty, anterior cruciate ligament reconstruction, and meniscus repair.

There is increasing interest in the technique called iPACK (infiltration between the popliteal artery and capsule of the knee), which involves injecting local anesthetics into the space between the popliteal artery and the posterior capsule of the knee. This approach blocks the terminal branches of the genicular nerves and the popliteal plexus, which innervate the posterior capsule of the knee, while sparing the main trunks of the tibial and common peroneal nerves. Therefore, the iPACK block appears advantageous by providing motor-sparing posterior knee analgesia with a lower likelihood of nerve or vascular injury under ultrasound guidance. Studies have shown that combining ACB with the iPACK block provides significantly better postoperative numerical rating scale (NRS) scores, knee range of motion, and ambulation distances compared to ACB alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with written informed consent
2. Patients over 18 years old undergoing elective total knee arthroplasty surgery
3. Patients with ASA I-II-III
4. Patients receiving spinal anesthesia

Exclusion Criteria:

1. Revision knee arthroplasty and bilateral total knee arthroplasty
2. Liver or kidney failure
3. Patients under 18 years old
4. Patients receiving general anesthesia
5. Allergy or intolerance to study medications
6. Body mass index (BMI) > 40 kg/m²
7. Chronic use of gabapentin/pregabalin (regular use for more than 3 months)
8. Chronic opioid use (opioid use for more than 3 months or daily oral morphine equivalent > 5 mg/day for 1 month)
9. Patients with ASA IV and those undergoing emergency surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Once eligibility is confirmed, patients will receive complete oral and written information about the study. Informed consent will be obtained before randomization and study-specific procedures.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the comparison of discharge times between patients undergoing total knee arthroplasty who receive an adductor canal block with and without the addition of an iPACK block. | Until discharge after surgery(Up to 6 days after the surgery)
  Total Knee Arthroplasty surgery results in shorter hospital stays

SECONDARY OUTCOMES:
The secondary outcome will be the assessment of whether the addition of an iPACK block to the adductor canal block reduces postoperative opioid consumption and pain scores by 50%, which will be considered significant. | Acute pain will be assessed after surgery until discharge(Up to 6 days after the surgery)
  İt is a pain intensity determination system based on the system where there person tells a point between 0=(no pain) 10=( unbearable pain) and to describe their pain

CONTACTS AND LOCATIONS:
Overall Officials: MURAT DEMİRCİOGLU, Study Chair — muratdemircioglu01@gmail.com
Locations (1):
- Murat Demircioglu, Aydin, Turkey (Türkiye)